CLINICAL TRIAL: NCT02199678
Title: A Randomized,Double Blind, Parallel Group, Placebo Controlled Dose Ranging Study to Assess the Analgesic Efficacy, Tolerability, Safety and Pharmacokinetic/Pharmacodynamic Properties of a Sublingual Wafer Formulation of Ketamine Following Third Molar Extraction
Brief Title: A Study to Assess the Analgesic Properties of a Sublingual Wafer Formulation of Ketamine Following Third Molar Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lotus Clinical Research, LLC (Other)
Collaborators: iX Biopharma Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KET003
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- ketamine 25 mg (Active Comparator): ketamine
  Interventions: Drug: ketamine 25 mg
- ketamine 35 mg (Active Comparator): ketamine
  Interventions: Drug: ketamine 35 mg
- ketamine 50 mg (Active Comparator): ketamine
  Interventions: Drug: ketamine 50 mg

INTERVENTIONS:
Drug: Placebo — placebo
  Arms: Placebo
Drug: ketamine 25 mg — ketamine
  Arms: ketamine 25 mg
Drug: ketamine 35 mg — ketamine
  Arms: ketamine 35 mg
Drug: ketamine 50 mg — ketamine
  Arms: ketamine 50 mg

SUMMARY:
This is a Phase 2, randomized, multicenter, parallel group, double-blind, dose-ranging, placebo-controlled evaluation of the analgesic efficacy, safety and pharmacokinetics of ketamine sublingual wafer in adult subjects who experience post operative pain after undergoing third molar extraction.

ELIGIBILITY:
18- 38 years of age Scheduled to undergo two ipsilateral third molar extractions

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Sum of Pain Intensity Difference | 3 hours
  The primary objective of this study is to demonstrate the dose-response relationship for analgesia of three dose levels of ketamine sublingual wafer compared with placebo, using the summed pain intensity difference from baseline over the first 3 hours (SPID3) in subjects with acute moderate to severe pain following third molar extraction.

SECONDARY OUTCOMES:
Sum of Pain Intensity Difference | 6 hours
  SPID 6
Safety and tolerability | 6 hours
  Safety and tolerability of ketamine sublingual wafer as evaluated with physical examination, vital signs, pulse oximetry, clinical laboratory tests, ECGs, and incidence of Adverse Events (AEs) and Serious AEs (SAEs)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lotus Clinical Research, LLC, Pasadena, California
  - Prahealthsciences, Salt Lake City, Utah